CLINICAL TRIAL: NCT04968002
Title: Application of Pablizumab Combined With Apatinib and Chemotherapy in Resectable Non-small Cell Lung Cancer： A Prospective, Single Arm, Single Center Phase II Clinical Study of Neoadjuvant Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0309
Record Dates: First submitted 2021-06-24; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Pabolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative neoadjuvant therapy for patients with stage IIa-IIIa non-small cell lung cancer. (Experimental): No EGFR mutation or ALK gene translocation was found in the untreated patients with NSCLC stage IIa-IIIb diagnosed by imaging, histopathology or cytology. After informed consent is signed by the patients. The patients were treated according to the protocols.
  Interventions: Drug: pablizumab combined with apatinib and neoadjuvant chemotherapy

INTERVENTIONS:
Drug: pablizumab combined with apatinib and neoadjuvant chemotherapy — The patients with stage IIa-IIIa non-small cell lung cancer are treated with pablizumab combined with apatinib and neoadjuvant chemotherapy

SUMMARY:
This is a prospective, single arm, single center clinical study to determine the efficacy and safety of pablizumab combined with apatinib and neoadjuvant chemotherapy in patients with stage iia-iiia non-small cell lung cancer. No EGFR mutation or ALK gene translocation was found in the untreated patients with NSCLC stage IIa-IIIb diagnosed by imaging, histopathology or cytology. After informed consent is signed by the patients. The patients were treated according to the protocols. The patients were followed up from adjuvant treatment and follow-up to relapse free survival until disease progression, withdrawal of informed consent, loss of follow-up or death.

ELIGIBILITY:
Inclusion Criteria:1. Age: 18-75 years old, male or female;

2. Non small cell lung cancer was diagnosed by imaging, histopathology or cytology

The resectable clinical stage assessed by the investigators was stage IIA - IIIA (according to AJCC)

TNM staging, 8th Edition);

3. ECoG PS score: 0-1;

4. According to the RECIST version 1.1 evaluation standard, at least one image can be measured

The lesions were measured;

5. There was no operation contraindication in preoperative organ function examination;

6. The laboratory examination indexes meet the requirements:

7. No previous treatment for NSCLC, including surgery and chemotherapy

Therapy, radiotherapy, targeted therapy, hormone or immunotherapy, etc;

8. Women of childbearing age agreed to use contraception during the study and within 6 months after the end of the study; study

The serum or urine pregnancy test was negative in the first seven days, and the patients were not in lactation

9. The subjects can understand the research situation and sign the informed consent voluntarily.

-

Exclusion Criteria: 1. Have received any treatment including chemotherapy in the past

Or radiotherapy;

2. The tumor has invaded important blood vessels or the tumor is in the treatment stage according to the judgment of the researcher

There is a high possibility of invading important blood vessels and causing massive hemorrhage;

3. Known EGFR mutation or ALK gene translocation;

4. There are locally advanced unresectable diseases and metastatic diseases;

5. She had been suffering from the need to use corticosteroids (prednisolone) in 14 days before randomization

Daily dose of nisone or equivalent (10 mg) or other immunosuppressive drugs

Any disease requiring systemic treatment. Local replacement steroids are permitted

(daily dose ≤ 10 mg of prednisone or equivalent) and prescription corticosteroids

Short term (≤ 7 days) prophylactic use of alcohol or for the treatment of non autoimmune.

Any active autoimmune disease or history of autoimmunity;

6. Active autoimmune diseases or autoimmune diseases that may recur

History. Admission of well controlled type I diabetes and hormone replacement therapy are allowed.

Hypothyroidism, well controlled celiac disease, and no need for complete treatment

Skin diseases (such as vitiligo, psoriasis or alopecia) treated by the body or not

Due to the absence of recurrence of the disease is not expected.

7. Interstitial lung disease, non infectious pneumonia or poorly controlled diseases (including pulmonary fibrosis)

History of vitamin C, acute lung disease, etc.

8. active hepatitis B (defined as screening hepatitis B virus surface antigen [HBsAg])

The results were positive and HBV-DNA was detected. The detection value was higher than that in the study

Upper limit of normal value of cardiology laboratory) or hepatitis C (defined as screening hepatitis C virus table)

The subjects with positive results of hcsab and HCV-RNA;

9. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive);

10. Inoculate live vaccine within 30 days before the first administration. Including but not limited to the following:

Mumps, rubella, measles, varicella / herpes zoster (varicella), yellow fever

Rabies, BCG and typhoid vaccine (inactivated virus vaccine allowed);

11. Suffering from uncontrolled clinical symptoms or diseases of the heart;

12. Long term antiplatelet therapy is needed;

13. Those who are allergic to any drug in this program;

14. Pregnant or lactating women;

15. According to the judgment of the researcher, the subjects may confuse the test results and interfere

It is not in the best interests of the subjects to participate in the whole trial

A history or current evidence of any disease, treatment, or laboratory abnormality

It's a good idea.

16. Active bleeding.

Exclusion criterion:

1. Ever received any treatment including chemotherapy or radiotherapy in the past;
2. The tumor has invaded important blood vessels. There is a high possibility of invading important blood vessels and causing massive hemorrhage if the tumor is in the treatment stage process according to the judgment of the researcher;
3. EGFR mutation or ALK gene translocation;
4. There are locally advanced unresectable diseases and metastatic diseases;
5. Patients had been suffering from the need to use corticosteroids (prednisolone) in 14 days before randomization grouping. Daily dose of nisone or equivalent (10 mg) or other immunosuppressive drugs. Any active autoimmune disease or history of autoimmunity;
6. Active autoimmune diseases or autoimmune diseases that may recur
7. Interstitial lung disease, non infectious pneumonia or poorly controlled diseases (including pulmonary fibrosis) etc.
8. active hepatitis B (defined as screening hepatitis B virus surface antigen [HBsAg]). And the results were positive and HBV-DNA was detected. The detection value was higher than that in the study upper limit of normal value of cardiology laboratory) or hepatitis C (defined as screening hepatitis C virus table and the subjects with positive results of hcsab and HCV-RNA;
9. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive);
10. Inoculated live vaccine within 30 days before the first administration. Including but not limited to the following: Mumps, rubella, measles, varicella / herpes zoster (varicella), yellow fever Rabies, BCG and typhoid vaccine (inactivated virus vaccine allowed);
11. Suffering from uncontrolled clinical symptoms or diseases of the heart;
12. Long term antiplatelet therapy is needed;
13. Those who are allergic to any drug in this program;
14. Pregnant or lactating women.;
15. According to the judgment of the researcher, the subjects may confuse and interfere the test results. It is not in the best interests of the subjects to participate in the whole trial.
16. Active bleeding patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The main pathological response rate | through surgical treatment completion, an average of 4 months
  After neoadjuvant therapy, the residual tumor was observed under microscope with a result of the proportion of tumor cells was less than or equal to 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China